CLINICAL TRIAL: NCT01092078
Title: Community-based Approaches to Treating Hypertension and Colon Cancer Prevention
Acronym: MISTER-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Cornell University (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Joseph E. Ravenell, MD, MS, Assistant Professor, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 09-0151
Record Dates: First submitted 2010-03-18; First posted 2010-03-24 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension; Colon Cancer
Keywords: hypertension; colon cancer screening; african american; men; motivational interviewing; patient navigation
MeSH Terms: conditions — Hypertension; Colonic Neoplasms; Multiple Endocrine Neoplasia Type 1 | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Motivational Interviewing (Experimental): Individuals in the motivational interviewing (MINT) arm of the study will receive telephone-based lifestyle interviewing for 6-months. Counseling will be aimed at modifying diet and/or physical activity behaviors associated with decreasing blood pressure.
  Interventions: Behavioral: MINT
- Patient Navigation (Experimental): Participants in the patient navigation arm will receive patient navigation for colonoscopy.
  Interventions: Behavioral: Patient Navigation
- PLUS (Experimental): Both patient navigation for colorectal cancer screening and motivational interviewing for blood pressure control
  Interventions: Behavioral: MINT; Behavioral: Patient Navigation

INTERVENTIONS:
Behavioral: MINT — Motivational interviewing for lifestyle changes associated with treating hypertension
  Arms: Motivational Interviewing; PLUS
Behavioral: Patient Navigation — Patient navigation for colonoscopy.
  Arms: PLUS; Patient Navigation

SUMMARY:
Black men constitute the demographic group with the greatest burden of premature death and disability from hypertension (HTN) in the United States. But while the disproportionately high rate of hypertension-related morbidity and mortality is well documented, the epidemic of colorectal cancer (CRC) among black men is comparatively under-appreciated. For example, CRC is a leading cause of cancer death in black men with a death rate 50% higher than in white men. Low rates of screening for CRC in this population contribute significantly to this problem. The purpose of this randomized controlled trial (RCT) is to evaluate the effect of a lifestyle intervention delivered through telephone-based motivational interviewing (MINT) versus a patient navigation intervention on blood pressure reduction and CRC screening.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be age 50 years or older,
2. Self-identify as a black or African American male,
3. Have uncontrolled hypertension as defined by systolic blood pressure (SBP) > 135 mmHg or diastolic blood pressure (DBP) > 85 mmHg and SBP > 130 or DBP > 80 mmHg (in those with diabetes at the screening).

Exclusion Criteria:

1. Inability to comply with the study protocol (either self-selected or by indicating during screening that he could not complete all requested tasks).

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Actual)
Dates: Start 2010-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Outcome is measured at 6-month follow-up
  Three blood pressure measures and the average of the three measures will be obtained at baseline and 6-month follow-up using a Welch Allyn Vital Signs automated blood pressure monitor.
Colon Cancer Screening Behavior | The outcome will be measured at 6-month follow-up
  Whether or not the participant was screened for colon cancer between baseline and 6-month follow-up will be assessed using self-report and patient medical records.

SECONDARY OUTCOMES:
Medication Adherence | 6-month follow-up
  Medication adherence will be assessed using the 4-item Morisky Medication Adherence scale.
Physical Activity | 6-month follow-up
  Physical activity will be measured using the International Physical Activity Questionnaire (IPAQ).
Intrinsic Motivation to Exercise | 6-month Follow-up
  Intrinsic motivation will be assessed using a 17-item questionnaire.
Self-Efficacy (Exercise) | 6-month follow-up
  Self-efficacy related to exercise will be measured using a 12-iten questionnaire.
Dietary Intake | 6-month follow-up
  Dietary intake will be assessed using the Food Frequency Questionnaire.
Intrinsic Motivation (Diet) | 6-month follow-up
  Intrinsic motivation relating to diet will be assessed using a 17-item scale.
Self-efficacy (Diet) | 6-month follow-up
  Self-efficacy relating to diet will be assessed using a 10-item scale.
Facilitators and Barriers to obtaining a colonoscopy | 6-month follow-up
  Facilitators and barriers to obtaining a colonoscopy will be assessed using a self-reported scale.
Behavioral Intention relating to colon cancer screening | 6-month follow-up
  Behavioral intention to screen for colon cancer will be assessed using a self-reported scale.
Social Influence relating to colon cancer screening | 6-month follow-up
  Social influence relating to colon cancer screening will be assessed using a self-reported questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ravenell, MD, MS, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Ravenell J, Thompson H, Cole H, Plumhoff J, Cobb G, Afolabi L, Boutin-Foster C, Wells M, Scott M, Ogedegbe G. A novel community-based study to address disparities in hypertension and colorectal cancer: a study protocol for a randomized control trial. Trials. 2013 Sep 8;14:287. doi: 10.1186/1745-6215-14-287. PMID 24011142
- [Derived] Cole H, Thompson HS, White M, Browne R, Trinh-Shevrin C, Braithwaite S, Fiscella K, Boutin-Foster C, Ravenell J. Community-Based, Preclinical Patient Navigation for Colorectal Cancer Screening Among Older Black Men Recruited From Barbershops: The MISTER B Trial. Am J Public Health. 2017 Sep;107(9):1433-1440. doi: 10.2105/AJPH.2017.303885. Epub 2017 Jul 20. PMID 28727540